CLINICAL TRIAL: NCT03064633
Title: Dexamethasone Versus Dexmedetomidine as Local Anesthetic Adjuvants in Ultrasound Guided Transversus Abdominis Plane Block for Total Abdominal Hysterectomies
Brief Title: Dexamethasone Versus Dexmedetomidine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fayoum University Hospital (Other)
Responsible Party: Principal Investigator, Hany Mahmoud Yassin, Dr., Fayoum University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M88
Record Dates: First submitted 2017-02-06; First posted 2017-02-27 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Postoperative Pain
Keywords: Dexamethasone; Dexmedetomidine; Transversus abdominis plane block; Local anesthetic adjuvants; postoperative pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Dexamethasone; Dexmedetomidine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexamethasone arm (group A) (Active Comparator): The local anesthetic solution mixture consists of dexamethasone 8 mg in Bupivacaine 0.25% Injectable Solution to a total volume of 40 ml (19 ml bupivacaine 0.5 % + 19 ml normal saline + 2 ml dexamethasone = 40ml). 20 ml of the local anesthetic solution mixture will be injected on each side.The Transversus abdominis Plane (TAP) block will be performed once after induction of anesthesia.
  Interventions: Drug: dexamethasone 8 mg; Drug: Bupivacaine 0.25% Injectable Solution
- Dexmedetomidine arm (group B) (Active Comparator): The local anesthetic solution mixture consists of dexmedetomidine 80 µg in Bupivacaine 0.25% Injectable Solution to a total volume of 40 ml (19 ml bupivacaine 0.5 % + 19 ml normal saline + 80 µg dexmedetomidine in 2 ml = 40ml). 20 ml of the local anesthetic solution mixture will be injected on each side.The Transversus abdominis Plane (TAP) block will be performed once after induction of anesthesia.
  Interventions: Drug: dexmedetomidine 80 µg; Drug: Bupivacaine 0.25% Injectable Solution

INTERVENTIONS:
Drug: dexamethasone 8 mg — At the level of the umbilicus, the high-frequency ultrasound linear array probe (L 4 - 12) will be placed transversely on the anterolateral abdominal wall between the subcostal margin and the iliac crest. localization of the fascial plane between the internal oblique and the transversus abdominis muscles will be done. The local anesthetic solution mixture will be injected with short bevel needle. The TAP block will be performed on the both side using the same technique and the same local anesthetic solution mixture volume. For the patients randomized to dexamethasone group, the local anesthetic solution mixture will consist of a total volume of 40 ml containing bupivacaine 0.25 % and dexamethasone 8 mg.
  Other Names: Dexamethasone 4 mg/ml
  Arms: Dexamethasone arm (group A)
Drug: dexmedetomidine 80 µg — At the level of the umbilicus, the high-frequency ultrasound linear array probe (L 4 - 12) will be placed transversely on the anterolateral abdominal wall between the subcostal margin and the iliac crest. localization of the fascial plane between the internal oblique and the transversus abdominis muscles will be done. The local anesthetic solution mixture will be injected with short bevel needle. The TAP block will be performed on the both sides using the same technique and the same local anesthetic solution mixture volume. For the patients randomized to dexmedetomidine group, the local anesthetic solution mixture will consist of a total volume of 40 ml containing bupivacaine 0.25 % and dexmedetomidine 80 µg.
  Other Names: precedex 100 µg/ml
  Arms: Dexmedetomidine arm (group B)
Drug: Bupivacaine 0.25% Injectable Solution — 38 ml of the solution will be prepared to be used in transversus abdominis plane block
  Other Names: Marcaine 0.25%

SUMMARY:
The transversus abdominis plane (TAP) block is most often used to provide surgical anesthesia for minor, superficial procedures on the lower abdominal wall, or postoperative analgesia for procedures below the umbilicus providing anesthesia to the ipsilateral lower abdomen below the umbilicus.

In a recent meta-analysis, the TAP block was shown to reduce the need for postoperative opioid use, increase the time to the first request for further analgesia, and provide more effective pain relief, while decreasing opioid-related side effects such as sedation and postoperative nausea and vomiting. The provision of effective postoperative analgesia is of key importance to facilitate early ambulation and prevention of postoperative morbidity. The analgesic regimen needs to meet the goals of providing safe, effective analgesia, with minimal side effects. Many additives to local anesthetics used to prolong the duration of analgesia for peripheral nerve blocks have been studied as dexamethasone, dexmedetomidine Dexmedetomidine is a lipophilic α2 agonist derivative with a higher affinity for α2-receptors than clonidine (α2: α1 specificity ratio is 200:1 for clonidine and 1600:1 for dexmedetomidine). It has sedative, analgesic, and sympatholytic effects that blunt many of the cardiovascular responses seen during the perioperative period. Animal and human studies have shown safety and efficacy of adding dexmedetomidine to local anesthetics in various regional anesthetic procedures. The addition of dexmedetomidine to bupivacaine in TAP block achieves better local anesthesia and provides better pain control postoperatively without any major side-effects.

Dexamethasone is a systemic glucocorticoid that improves the quality of recovery after surgery by reducing pain, nausea, and vomiting. When added to local anesthetics as an adjuvant in peripheral blocks, it prolongs the analgesia time. Mechanism of action may be through the anti-inflammatory action, the increase of the local efficiency, and to slow down of the absorption.

Objective:

The objective is to compare and evaluate efficacy and safety of dexmedetomidine and dexamethasone as a local anesthetic adjuvant to bupivacaine in ultrasound-guided TAP block for patients scheduled for total abdominal hysterectomies.

DETAILED DESCRIPTION:
PATIENTS AND METHODS:

This study will be performed on Fifty-four adult patients who will be undergone an abdominal hysterectomy after obtaining the approval of the local ethical committee and scientific institutional review board. written informed consents will be signed from each patient before enrollment and randomization into the study.

The patients will be randomly allocated to receive either a mixture of bupivacaine and dexamethasone 8 mg (group A, 27 patients) or a mixture of bupivacaine and dexmedetomidine 80 µg (group B, 27 patients). Randomization will be performed by using a computer-generated random number list. The random number for each patient will be concealed in opaque sealed envelope which will be opened by the investigators shortly after the admission of the patient into the operation room. The investigators sharing in the patients care and data acquisition will be blinded to groups allocation till full completion of statistical analysis.

Preoperative preparation:

Visual analog scale (VAS) will be explained to all the patients on preoperative visit (0-10 cm, in which 0 cm = no pain and 10 cm = worst pain) and the compulsory investigations according to the regular institutional protocol will be done [electrocardiogram (ECG), complete blood count (CBC), blood sugar level, serum urea and creatinine, liver function tests, and coagulation profile].

On the day of surgery, intravenous (IV) access will be inserted. The patient will be administered midazolam 0.03 mg/kg, metoclopramide 10 mg slowly, ranitidine 50 mg, and cefotaxime 1 gm intravenously (IV) as premedications.

Anesthetic technique:

All the patients will be received a standard general anesthesia with standard monitoring [ECG, noninvasive blood pressure (NIBP), capnography and pulse oximetry]. Anesthesia will be induced by using fentanyl 1μg/kg, propofol 1.5-2 mg/kg and Atracurium 0.5 mg/kg will be used for muscle relaxation to facilitate endotracheal intubation by cuffed endotracheal tube (internal diameter = 7 mm).

After induction of anesthesia and under a complete aseptic condition, the TAP blocks will be performed by the attending anesthesiologists who will not participate in this trial under real-time ultrasound guidance (Philips ClearVue 350 Ultrasound Machine, Philips healthcare, USA). At the level of the umbilicus, the high-frequency ultrasound linear array probe (L4 - 12) will be placed transversely on the anterolateral abdominal wall between the subcostal margin and the iliac crest. Identification of the external oblique, the internal oblique, and the transversus abdominis muscles and localization of the fascial plane between the internal oblique and the transversus abdominis muscle that appeared as a hypoechoic line will be done. The local anesthetic solution mixture will be injected with short bevel needle (22 Gauge, 90 mm sonoplex stim cannula, Pajunk® GmbH, Geisingen, Germany) under real-time ultrasound guidance after negative aspiration to avoid intravascular injection. The local anesthetic solution mixture will be observed separating the fascial plane during injection. The TAP block will be then performed on the opposite side, using the same technique and the same local anesthetic solution mixture volume. For the patients randomized to group A (dexamethasone group, 27 patients), the local anesthetic solution mixture consisted of a total volume of 40 ml bupivacaine 0.25 % and dexamethasone 8 mg, 20 ml injected on each side. Dexamethasone sodium phosphate (Epidron®, EIPICO, Cairo, Egypt) is supplied in 4 mg/ml ampule. For the patients randomized to group B (dexmedetomidine group, 27 patients), the local anesthetic solution mixture consisted of a total volume of 40 ml bupivacaine 0.25 % and dexmedetomidine 80 µg, 20 ml injected on each side. Dexmedetomidine hydrochloride (Precedex®, manufactured by Hospira, Inc. Lake Forest, IL, and USA) is supplied in 100 μg/ml ampule. the local anesthetic solution mixture will be prepared and coded by independent attending anesthesiologists who will not share in data collection or in patients care.

Anesthesia will be maintained with isoflurane 1.5 volume % and Atracurium 0.1 mg/kg will be administered as a maintenance dose every 30 minutes until completion of the procedure. Ventilation parameters will be adjusted as follows: tidal volume (TV) = 4-8 ml/kg, positive end-expiratory pressure (PEEP) = 5 cm H2O, respiratory rate (RR) = 12/min then it will be adjusted to maintain end-tidal CO2 between 35-40 mmHg, and fraction of inspired oxygen (FiO2) = 0.5-0.6.

Fentanyl 0.5μg/kg will be given intraoperatively when either heart rate or NIBP increased by more than 20% of the basal records and could be repeated till the desired effect. After completion of the procedure, anesthesia will be discontinued and tracheal extubation will be done once the extubation criteria will be fulfilled. The patients then will be transferred to the post-anesthesia care unit (PACU) for two hours' observation period. The patients will be discharged to the ward after fulfilling the discharge criteria based on modified Aldrete score ≥ 9.(17) As a part of standardized regular institutional postoperative pain control policy, Acetaminophen 1 gm every 6 hours by IV infusion and ketorolac 30 mg diluted in 100 ml normal saline through IV infusion over 20 minutes every 8 hours will be administered. Patients with VAS ≥ 5 received morphine sulfate IV at a bolus dose of 2-5 mg increments with a maximum dose of 15 mg per 4 hours or 45 mg per 24 hours. The criteria to stop morphine titration will be reasonable pain control or the patient became sedated (Ramsay sedation scale >2). Furthermore, respiratory rate < 10 / min, Oxygen saturation < 95%, or development of serious adverse effects (allergy, marked itching, excessive vomiting, and hypotension with systolic blood pressure ≤ 20% of baseline readings).

STATISTICAL ANALYSIS:

The normally distributed numerical data will be presented as mean (SD) and differences between groups will be compared using Student's t-tests. Continuous data with skewness and kurtosis as well as the ordinal data will be presented as median (interquartile range[IQR]) and compared for significance by using the Mann-Whit¬ney U test. The Kolmogorov-Smirnov test will be implemented to check the normality of Continuous data distribution (P ≤ 0.05). Categorical data will be presented as proportions and will be compared for significance by using the chi-square test. Fisher's exact test will be used instead if the minimum expected cell count less than five. We will use the log-rank test and Kaplan-Meier curves to compare data measuring time to an event. The level P ≤ 0.05 will be considered the cut-off value for significance. Statistical analysis will be performed using the statistical package for the social sciences (SPSS) version 16 (SPSS Inc., Chicago, IL, USA).

The sample size of 22 patients per group was found acceptable to detect a difference of 65 minutes between both groups in time for the first request of analgesia (primary outcome), assuming α = 0.05 (two tail), β = 0.2 (80 % power), and the standard deviation = 75 minutes (derived from Ammar et al. 2012). Recruitment of 27 patients per group will be done to account for possible data loss. Sample size calculation will be done by using G*Power software version 3.1.9.2 (Institute of Experimental Psychology, Heinrich Heine University, Dusseldorf, Germany).

ELIGIBILITY:
Inclusion Criteria:

* American society of anesthesiologists (ASA) physical status grade 1 and 2.
* Age of 18 years and more.
* Patients who will be scheduled for total abdominal hysterectomies.

Exclusion Criteria:

* Patient refusal.
* Body mass index (BMI) > 40.
* Patients with chronic pain and those using chronic analgesic medications.
* Coagulopathy.
* Allergy to the study drugs.
* Patients taking other medications with α-adrenergic blocking effect.
* Hepatic or renal insufficiency.
* Systemic infection.
* Infection at the site of injection.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2017-03-08 (Actual); Primary Completion 2018-04-28 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Time to first request of analgesia | During the 24 hours postoperatively
  The time passed till the patient request an analgesic dose

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) at rest | Assesment will be done at 2 hours postoperatively
  Range from 0-10 cm, in which 0 cm=no pain and 10 cm=worst pain
Visual Analog Scale (VAS) at rest | Assesment will be done at 4 hours postoperatively
  Range from 0-10 cm, in which 0 cm=no pain and 10 cm=worst pain
Visual Analog Scale (VAS) at rest | Assesment will be done at 6 hours postoperatively
  Range from 0-10 cm, in which 0 cm=no pain and 10 cm=worst pain
Visual Analog Scale (VAS) at rest | Assesment will be done at 12 hours postoperatively
  Range from 0-10 cm, in which 0 cm=no pain and 10 cm=worst pain
Visual Analog Scale (VAS) at rest | Assesment will be done at 18 hours postoperatively
  Range from 0-10 cm, in which 0 cm=no pain and 10 cm=worst pain
Visual Analog Scale (VAS) at rest | Assesment will be done at 24 hours postoperatively
  Range from 0-10 cm, in which 0 cm=no pain and 10 cm=worst pain
Visual Analog Scale (VAS) at rest | Assesment will be done at 48 hours postoperatively
  Range from 0-10 cm, in which 0 cm=no pain and 10 cm=worst pain
Visual Analog Scale (VAS) on movement | Assesment will be done at 2 hours postoperatively
  Range from 0-10 cm, in which 0 cm=no pain and 10 cm=worst pain
Visual Analog Scale (VAS) on movement | Assesment will be done at 4 hours postoperatively
  Range from 0-10 cm, in which 0 cm=no pain and 10 cm=worst pain
Visual Analog Scale (VAS) on movement | Assesment will be done at 6 hours postoperatively
  Range from 0-10 cm, in which 0 cm=no pain and 10 cm=worst pain
Visual Analog Scale (VAS) on movement | Assesment will be done at 12 hours postoperatively
  Range from 0-10 cm, in which 0 cm=no pain and 10 cm=worst pain
Visual Analog Scale (VAS) on movement | Assesment will be done at 18 hours postoperatively
  Range from 0-10 cm, in which 0 cm=no pain and 10 cm=worst pain
Visual Analog Scale (VAS) on movement | Assesment will be done at 24 hours postoperatively
  Range from 0-10 cm, in which 0 cm=no pain and 10 cm=worst pain
Visual Analog Scale (VAS) on movement | Assesment will be done at 48 hours postoperatively
  Range from 0-10 cm, in which 0 cm=no pain and 10 cm=worst pain
Interval doses of consumed morphia | During 0 - 2 hours postoperatively
  Morphine doses consumed at different times
Interval doses of consumed morphia | During 2 - 4 hours postoperatively
  Morphine doses consumed at different times
Interval doses of consumed morphia | During 4 - 6 hours postoperatively
  Morphine doses consumed at different times
Interval doses of consumed morphia | During 6 - 12 hours postoperatively
  Morphine doses consumed at different times
Interval doses of consumed morphia | During 12 - 18 hours postoperatively
  Morphine doses consumed at different times
Interval doses of consumed morphia | During 18 - 24 hours postoperatively
  Morphine doses consumed at different times
Interval doses of consumed morphia | During 24 - 48 hours postoperatively
  Morphine doses consumed at different times
Cumulative doses of consumed morphia | During the 24 hours postoperatively
  Total morphine doses consumed during the 24 hours postoperatively.
Intraoperative fentanyl consumption | At the end of surgical procedure
  total doses of fentanyl consumed during the surgical procedure intraoperatively.
Nausea | During the 48 hour postoperatively
  incidence of nausea
Vomiting | During the 48 hour postoperatively
  incidence of vomiting
Sedation score | At 2 hours postoperatively
  Degree of sedation: where:1= Fully awake and oriented, 2= Drowsy, 3= Eye closed but responds to commands, 4= Eye closed but responds to mild physical stimulation, 5= Eye closed and not responding to mild physical stimulation
Sedation score | At 4 hours postoperatively
  Degree of sedation: where:1= Fully awake and oriented, 2= Drowsy, 3= Eye closed but responds to commands, 4= Eye closed but responds to mild physical stimulation, 5= Eye closed and not responding to mild physical stimulation
Sedation score | At 6 hours postoperatively
  Degree of sedation: where:1= Fully awake and oriented, 2= Drowsy, 3= Eye closed but responds to commands, 4= Eye closed but responds to mild physical stimulation, 5= Eye closed and not responding to mild physical stimulation
Sedation score | At 12 hours postoperatively
  Degree of sedation: where:1= Fully awake and oriented, 2= Drowsy, 3= Eye closed but responds to commands, 4= Eye closed but responds to mild physical stimulation, 5= Eye closed and not responding to mild physical stimulation
Sedation score | At 18 hours postoperatively
  Degree of sedation: where:1= Fully awake and oriented, 2= Drowsy, 3= Eye closed but responds to commands, 4= Eye closed but responds to mild physical stimulation, 5= Eye closed and not responding to mild physical stimulation
Sedation score | At 24 hours postoperatively
  Degree of sedation: where:1= Fully awake and oriented, 2= Drowsy, 3= Eye closed but responds to commands, 4= Eye closed but responds to mild physical stimulation, 5= Eye closed and not responding to mild physical stimulation
Sedation score | At 48 hours postoperatively
  Degree of sedation: where:1= Fully awake and oriented, 2= Drowsy, 3= Eye closed but responds to commands, 4= Eye closed but responds to mild physical stimulation, 5= Eye closed and not responding to mild physical stimulation
Hypotension | During intraoperative period
  incidence of hypotension (systolic blood pressure < 90 mmHg)
Hypotension | During 48 hours postoperatively
  incidence of hypotension (systolic blood pressure < 90 mmHg)
Bradycardia | During intraoperative period
  Incidence of bradycardia ( heart rate < 60 beat/minute)
Bradycardia | During 48 hours postoperatively
  Incidence of bradycardia ( heart rate < 60 beat/minute)

CONTACTS AND LOCATIONS:
Overall Officials: Hany M Yassin, MD, Principal Investigator — Fayoum University Hospital
Locations (1):
- Fayoum University hospital, El Fayoum Qesm, Faiyum Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ammar AS, Mahmoud KM. Effect of adding dexamethasone to bupivacaine on transversus abdominis plane block for abdominal hysterectomy: A prospective randomized controlled trial. Saudi J Anaesth. 2012 Jul;6(3):229-33. doi: 10.4103/1658-354X.101213. PMID 23162395
- [Background] Almarakbi WA, Kaki AM. Addition of dexmedetomidine to bupivacaine in transversus abdominis plane block potentiates post-operative pain relief among abdominal hysterectomy patients: A prospective randomized controlled trial. Saudi J Anaesth. 2014 Apr;8(2):161-6. doi: 10.4103/1658-354X.130683. PMID 24843325
- [Background] Abdallah FW, Brull R. Facilitatory effects of perineural dexmedetomidine on neuraxial and peripheral nerve block: a systematic review and meta-analysis. Br J Anaesth. 2013 Jun;110(6):915-25. doi: 10.1093/bja/aet066. Epub 2013 Apr 15. PMID 23587874
- [Background] Gadsden J, Ayad S, Gonzales JJ, Mehta J, Boublik J, Hutchins J. Evolution of transversus abdominis plane infiltration techniques for postsurgical analgesia following abdominal surgeries. Local Reg Anesth. 2015 Dec 10;8:113-7. doi: 10.2147/LRA.S96253. eCollection 2015. PMID 26677342